CLINICAL TRIAL: NCT00507754
Title: Latent Mycobacterium Tuberculosis Infection Among Cancer Patients
Brief Title: Latent Tuberculosis Infection in Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1095
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Solid Tumors; Latent Mycobacterium Tuberculosis; Tuberculin Skin Test; Tuberculosis; T-SPOT TB test; TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample will be collected and used to perform the T-SPOT. TB test.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Latent Tuberculosis Infection: Patients with cancer at risk for developing active tuberculosis (TB).
  Interventions: Other: T-SPOT TB test

INTERVENTIONS:
Other: T-SPOT TB test — Extra blood draw, followed by ten minutes rest and the injection of Tuberculin subcutaneously on forearm.

SUMMARY:
Primary Objective:

1. To evaluate the performance of the new T-SPOT.TB test and the conventional TST for screening of Latent Tuberculosis infections in patients with cancer and those undergoing Hematopoietic Stem Cell Transplant.

Secondary Objectives:

1. To examine the factors associated with positive response to T-SPOT.TB and the TST (tuberculin skin test) in patients with anergy.
2. To determine the impact of immunosuppressive and antineoplastic therapy on the screening performance of T-SPOT.TB and the TST in cancer patients.

DETAILED DESCRIPTION:
TB AND TB TESTS:

Patients with cancer are considered "immunocompromised." This means that, because of the cancer and the cancer treatment, the immune system does not function normally, which decreases its ability to fight off infection and disease. This immunocompromised condition places these patients (who probably had been in contact with the TB bacteria, resulting in latent, or inactive, TB) at risk for active TB. Latent TB does not cause symptoms or signs of active TB infection. It is very important to identify patients who are at risk for developing active TB, so that they can receive timely treatment for TB.

The Tuberculin skin test (TST) is currently used to detect latent TB. The TST is considered to have low detection sensitivity, which means that it may not always detect latent TB, which may then turn into an active TB infection.

The T-SPOT.TB is a new test that researchers want to study to see whether it may be more effective and accurate than the TST at identifying patients at risk for developing active TB.

STUDY PARTICIPATION:

If you agree to take part in this study, you will have the following tests done and steps taken.

* You will have extra blood (about 1 to 2 teaspoons) drawn. It will be done at the same time as your routine clinic visit to M. D. Anderson or as a regular blood draw if you are already admitted in the hospital. This blood will be used to perform the T-SPOT. TB test.

If you have had a TST (or tuberculin skin test) performed at M. D. Anderson in the past 45 days, it may probably not be necessary to repeat the TST. However, the research staff will decide if you need to have a new TST.

You may have the TST performed before or after your blood is drawn. In any case, you will rest for 10 minutes after the blood draw.

* You will receive a fluid called tuberculin in order to have the TST performed. Tuberculin will be injected just beneath the surface of the skin on your forearm. You should then see a very small raised area of skin where the injection was given. This reaction will wear off in a few days.
* After 2-3 days (48-72 hours later), you will return to M. D. Anderson (if you are not in the hospital), and a health care professional will look at and measure any swelling or redness at the site of TST. The doctor will then learn if your TST result is positive or negative. If your TST is positive the study doctor will discuss it with , your primary doctor for further evaluation and treatment.

Although you will be informed about the TST result, you will not be informed about the T-SPOT. TB test result because the T-SPOT. TB test is just used for investigational purposes in this study and will not be used for diagnostic purposes. The study doctor will use the results of the T-SPOT. TB test to make research comparisons with the TST test results.

LENGTH OF STUDY:

Your participation will be over in this study once both TB tests have been performed and the TST has been checked by a health care professional.

This is an investigational study. The TST is FDA approved and commercially available. The T-SPOT.TB test is not FDA approved or commercially available. It is authorized for use in research only. Up to 200 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* Patients who are receiving chemotherapy for hematologic malignancy and solid-organ cancer.
* Patients with a Hematopoietic stem cell transplantation (HSCT) history will be included after >1 year of transplantation.

Exclusion Criteria:

* Refusal of consent
* Individuals who, on the advice of the Primary or enrolling physician, may otherwise be at increased risk of an adverse reaction to venipuncture or tuberculin skin test administration.
* Lymphocytopenia (< 300 cells/microliter)
* Patients with known HIV infection.
* Patients with known active tuberculosis will not be included in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with cancer at risk for developing active tuberculosis (TB).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Rate of Positive Results of T-SPOT.TB (%) | Study period 2 Years
  Number participants with postitive T-SPOT.TB test results compared to total positive results, derived from Center for Disease Control (CDC) Criteria used for LTBI positive skin test (i.e. a tuberculin skin test (TST) with 5 mm or more of induration). For those individuals with >5 mm induration on TST, chest radiograph performed. Fisher's exact test used to assess the association between categorical variables and the testing results of T-SPOT.TB or TST.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Safdar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org